CLINICAL TRIAL: NCT00412113
Title: A 6-Week, Prospective, Randomized, Double-Blind, Double-Dummy Phase IV Clinical Trial Designed to Evaluate the Efficacy of an Aggressive Multi-Risk Factor Management Strategy With Caduet (A3841045) Versus a Guideline-Based Approach in Achieving Blood Pressure and Lipid Goals in Hypertensive Subjects With Additional Risk Factors.
Brief Title: A Multi-Risk Factor Strategy vs a Guideline-Based Approach in Achieving Blood Pressure and Lipid Goals in Hypertensives at Extra Risk
Acronym: TOGETHER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3841045
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Results first posted 2009-11-06 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Dyslipidemia; Hypertension
MeSH Terms: conditions — Dyslipidemias; Hypertension | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Norvasc 5 mg (Active Comparator): Blinded amlodipine 5 mg and amlodipine/atorvastatin single pill combination 5/20 mg placebo dosed once daily for 6 weeks.
  Interventions: Drug: Amlodipine besylate
- Caduet 10/20mg (Experimental): Blinded amlodipine/atorvastatin single pill combination 10/20 mg dosed once daily for 6 weeks and amlodipine besylate 10 mg placebo.
  Interventions: Drug: Amlodipine besylate/atorvastatin calcium single pill combination
- Norvasc 10 mg (Active Comparator): Blinded amlodipine 19 mg and amlodipine/atorvastatin single pill combination 10/20 mg placebo dosed once daily for 6 weeks.
  Interventions: Drug: Amlodipine besylate
- Caduet 5/20mg (Experimental): Blinded amlodipine/atorvastatin single pill combination 5/20 mg and amlodipine besylate 5 mg placebo dosed once daily for 6 weeks .
  Interventions: Drug: Amlodipine besylate/atorvastatin calcium single pill combination

INTERVENTIONS:
Drug: Amlodipine besylate — Amlodipine besylate 5 mg
  Arms: Norvasc 5 mg
Drug: Amlodipine besylate/atorvastatin calcium single pill combination — Amlodipine/atorvastatin single pill combination 10/20 mg
  Arms: Caduet 10/20mg
Drug: Amlodipine besylate — Amlodipine besylate 10 mg
  Arms: Norvasc 10 mg
Drug: Amlodipine besylate/atorvastatin calcium single pill combination — Amlodipine/atorvastatin single pill combination 5/20 mg
  Arms: Caduet 5/20mg

SUMMARY:
The purpose of this study is to investigate whether an aggressive multi-risk factor management strategy (Caduet plus therapeutic lifestyle changes (TLC) regimen) will result in greater percentage of patients achieving blood pressure and low density lipoprotein cholesterol (LDL-C) goals compared with a Joint National Committee 7/ National Cholesterol Education Program Adult Treatment Panel III (JNC 7/NCEP ATP III) guideline-based approach (Norvasc plus TLC regimen) after 6 weeks of treatment in primary prevention subjects with hypertension and additional risk factors, including dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosed hypertension receiving treatment with Norvasc 5 or 10 mg and who also have 3 additional cardiovascular risk factors, including dyslipidemia.

Exclusion Criteria:

* Subjects who are taking the following prohibited medications within 14 days of screening: lipid-lowering therapy, calcium channel blocker other then Norvasc, >3 antihypertensive agents (including Norvasc)
* Subjects that have not been on a stable dose of Norvasc for at least 4 weeks
* Subjects with a history of coronary heart disease, stroke, or Pulmonary Vascular Disease (PVD)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (47):
- United States (47):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Garden Grove, California
  - Pfizer Investigational Site, Mission Viejo, California
  - Pfizer Investigational Site, Rancho Santa Margarita, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Safety Harbor, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Augusta, Georgia
  - Pfizer Investigational Site, Tucker, Georgia
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Erlanger, Kentucky
  - Pfizer Investigational Site, Auburn, Maine
  - Pfizer Investigational Site, Warren, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Chesterfield, Missouri
  - Pfizer Investigational Site, Florissant, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Belvidere, New Jersey
  - Pfizer Investigational Site, Bridgewater, New Jersey
  - Pfizer Investigational Site, Clifton, New Jersey
  - Pfizer Investigational Site, Elizabeth, New Jersey
  - Pfizer Investigational Site, Hillsborough, New Jersey
  - Pfizer Investigational Site, Trenton, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Lansdale, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Goose Creek, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Chesapeake, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841045&StudyName=A%20Multi-Risk%20Factor%20Strategy%20Vs%20A%20Guideline-Based%20Approach%20In%20Achieving%20Blood%20Pressure%20%26%20Lipid%20Goals%20In%20Hypertensives%20At%20Extra%20Risk

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled 244 evaluable subjects. Drug treatments were used prior to the start of the study in all subjects in the Caduet and therapeutic lifestyle changes (TLC) group and the Norvasc and TLC group. Amlodipine was used by all subjects prior to entry. The study's four arms are two groups, each with drug group and matching placebo.
Groups:
- Norvasc + TLC: Blinded Norvasc (amlodipine) 5 to 10 milligram (mg) and matching Caduet placebo dosed once daily along with Therapeutic Lifestyle Changes (TLC) for 6 weeks.
- Caduet + TLC: Blinded Caduet (amlodipine besylate/atorvastatin calcium) 5/20 to 10/20 mg and matching Norvasc placebo dosed once daily along with TLC for 6 weeks.
Period: Overall Study
Arm/Group | Norvasc + TLC | Caduet + TLC
Started | 123 (15-January-2007) | 122 (15-January-2007)
Received Treatment | 122 (One subject assigned to Norvasc and TLC did not receive treatment and was excluded from all analyses) | 122
Completed | 111 (15-April-2008) | 107 (15-April-2008)
Not Completed | 12 | 15
Not completed — Adverse Event | 11 | 15
Not completed — did not receive treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Norvasc + TLC | Caduet + TLC | Total
Number analyzed (Participants) | 122 | 122 | 244
Age, Customized [Number; unit: participants]
  18 to 64 years | 95 | 97 | 192
  > or = to 65 years | 27 | 25 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 65 | 121
  Male | 66 | 57 | 123

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Blood Pressure (BP) <140/90 Millimeters of Mercury (mmHg) and Low Density Lipoprotein Cholesterol (LDL-C) <100 Milligrams Per Deciliter(mg/dL) at Week 6
Description: Number of subjects reaching dual goal of systolic blood pressure <140 millimeters of mercury (mmHg) and diastolic blood pressue of <90 mmHg and low density lipoprotein-cholesterol(LDL-C) <100 milligrams per deciliter(mg/dL)
Time Frame: Week 6
Population: Full analysis set (FAS) is all randomized subjects who take at least one dose of study drug and and have any post-baseline efficacy assessments.
Measure: Number; unit: participants
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
participants | 11 | 80
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the percentage of patients achieving both the BP(< 140/90 mmHg) and LDL goal (< 100mg/dL) at Week 6. With ~120 in each treatment arm, planned power was at least 90% to detect a difference between treatments, assuming 35% in the Caduet and 15% in the Norvasc arm achieving BP <140/90 mmHg and LDL <100 mg/dL and using a chi-square test with 0.05 two-sided significance level; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — There was only one primary endpoint and the p-value was not adjusted for comparison; Odds Ratio (OR) = 19.03, 95% CI [9.14 to 39.63]

2. Secondary Outcome: Subjects With Blood Pressure of <140/90 mmHg and LDL-C <100 mg/dL at Week 4
Description: Subjects achieving both the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC)-7 blood pressure goal of <140/90 mmHg and the National Cholesterol Education Program Adult Treatment Panel (NCEP/ATP) III Update low density lipoprotein-cholesterol (LDL-C) goal <100 mg/dL at Week 4.
Time Frame: Week 4
Population: Full analysis set. All randomized subjects who took study drug and had at least one post-baseline efficacy assessment comprised the FAS.
Measure: Number; unit: participants
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 116
participants | 6 | 73
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the percentage of patients achieving both the blood pressure (< 140/90 mmHg) and LDL-goal (<100 mg/dL) at Week 4; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No adjustment for p-value for secondary analysis; Odds Ratio (OR) = 31.39, 95% CI [12.61 to 78.09]

3. Secondary Outcome: Subjects With BP <140/90 mmHg and LDL-C <130 mg/dL at Week 4.
Description: Subjects achieving both JNC-7 blood pressure goal of <140/90 mmHg and NCEP/ATP III LDL-C goal <130 mg/dL at Week 4.
Time Frame: Week 4
Population: Full analysis set (FAS). All randomized subjects who took study drug and had at least one post-baseline efficacy assessment comprised the FAS.
Measure: Number; unit: participants
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
participants | 41 | 85
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the percentage of patients achieving both the blood pressure (< 140/90 mmHg) and LDL-goal (<130mg/dL) at Week 4; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No adjustment for p-value for secondary analyses; Odds Ratio (OR) = 5.2, 95% CI [2.93 to 9.24]

4. Secondary Outcome: Subjects With BP <140/90 mmHg and LDL-C <130 mg/dL at Week 6.
Description: Subjects achieving both JNC-7 blood pressure goal of <140/90 mmHg and NCEP/ATP III LDL-C goal <130 mg/dL at Week 6.
Time Frame: Week 6
Population: Full analysis set (FAS).
Measure: Number; unit: participants
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
participants | 45 | 90
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the percentage of patients achieving both the blood pressure (< 140/90 mmHg) and LDL-goal (<130mg/dL) at Week 6; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No adjustment for p-value for secondary analyses; Odds Ratio (OR) = 5.14, 95% CI [2.89 to 9.11]

5. Secondary Outcome: Subjects With LDL-C < 100 mg/dL at Week 4
Description: Subjects Who achieve a goal of LDL-C < 100 mg/dL at Week 4.
Time Frame: Week 4
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
participants | 8 | 96
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the percentage of patients achieving (<100mg/DL) at Week 4; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No adjustment for p-value for secondary analyses; Odds Ratio (OR) = 65.51, 95% CI [27.10 to 158.34]

6. Secondary Outcome: Subjects With LDL-C < 100 mg/dL at Week 6
Description: Subjects Who achieve a goal of LDL-C < 100 mg/dL at Week 6.
Time Frame: Week 6
Population: Full analysis set (FAS) All randomized subjects who take at least one dose of study drug and have any post-baseline efficacy assessments.
Measure: Number; unit: participants
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
participants | 13 | 99
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the percentage of patients achieving LDL-goal (<100mg/DL) at Week 6; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No adjustment for p-value for secondary analyses; Odds Ratio (OR) = 42.04, 95% CI [19.42 to 90.99]

7. Secondary Outcome: Subjects With BP < 140/90 mmHg at Week 4
Description: Subjects achieving BP goal of <140/90 mmHg at week 4
Time Frame: Week 4
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 117
participants | 84 | 87
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the percentage of patients achieving blood pressure (< 140/90 mmHg)at Week 4; Test type: Superiority or Other; p = 0.785, Cochran-Mantel-Haenszel — No adjustment for p-value for secondary analyses; Odds Ratio (OR) = 1.09, 95% CI [0.60 to 1.98]

8. Secondary Outcome: Subjects With BP < 140/90 mmHg at Week 6
Description: Subjects achieving BP goal of <140/90 mmHg at week 6
Time Frame: Week 6
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
participants | 83 | 94
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the percentage of patients achieving blood pressure (< 140/90 mmHg) at Week 6; Test type: Superiority or Other; p = 0.171, Cochran-Mantel-Haenszel — No adjustment for p-value for secondary analyses; Odds Ratio (OR) = 1.55, 95% CI [0.83 to 2.88]

9. Secondary Outcome: Change From Baseline to Week 4 in Systolic Blood Pressure (SBP).
Description: Mean at observation minus mean at baseline
Time Frame: Week 4, baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mmHg | -2.6 (12.1) | -1.5 (11.9)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in systolic blood pressure at Week 4; Test type: Superiority or Other; p = 0.585, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = 0.76, 95% CI [-1.97 to 3.48]

10. Secondary Outcome: Change From Baseline to Week 4 in Diastolic Blood Pressure (DBP)
Description: Mean at observation minus mean at baseline
Time Frame: Week 4, baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mmHg | -1.5 (7.7) | -1.2 (8.8)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in diastolic blood pressure at Week 4; Test type: Superiority or Other; p > 0.999, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -0.00, 95% CI [-2.01 to 2.01]

11. Secondary Outcome: Change From Baseline to Week 4 in Pulse Rate
Description: Mean at observation minus mean at baseline measured in beats per minute (bpm).
Time Frame: Week 4, baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
bpm | -0.1 (8.2) | -0.9 (8.5)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in pulse rate at Week 4; Test type: Superiority or Other; p = 0.363, ANCOVA; Difference in LS Means = -0.90, 95% CI [-2.83 to 1.04]

12. Secondary Outcome: Change From Baseline to Week 6 in Systolic Blood Pressure (SBP)
Description: Mean change at observation minus mean baseline.
Time Frame: Week 6, baseline
Population: Full analysis set: all randomized subjects who take at least one dose of study drug and have any post-baseline efficacy assessments.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mmHg | -1.0 (12.6) | -4.0 (11.0)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in systolic blood pressure at Week 6; Test type: Superiority or Other; p = 0.020, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS means = -3.25, 95% CI [-5.99 to -0.51]

13. Secondary Outcome: Change From Baseline to Week 6 in Diastolic Blood Pressue (DBP)
Description: Change from mean at observation minus mean at baseline
Time Frame: Week 6, baseline
Population: as for outcome 3
Measure: Median (Standard Deviation); unit: mmHg
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mmHg | -1.1 (7.1) | -1.7 (8.2)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in diastolic blood pressure at Week 6; Test type: Superiority or Other; p = 0.351, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -0.87, 95% CI [-2.71 to 0.97]

14. Secondary Outcome: Change From Baseline to Week 6 in Pulse Rate
Description: Mean at observation minus mean at baseline
Time Frame: Week 6, baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
bpm | 0.9 (8.1) | 1.1 (9.0)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in mean change from baseline in pulse rate at Week 6; Test type: Superiority or Other; p = 0.922, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = 0.10, 95% CI [-1.91 to 2.11]

15. Secondary Outcome: Change From Baseline in LDL at Week 4.
Description: Change: mean of observation minus mean at baseline.
Time Frame: Week 4, baseline
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mg/dL | -0.5 (23.0) | -47.8 (24.4)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in LDL at Week 4; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -49.30, 95% CI [-54.68 to -43.91]

16. Secondary Outcome: Change From Baseline in High Density Lipoprotein (HDL) at Week 4.
Description: Mean change at observation minus baseline.
Time Frame: Week 4, baseline
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mg/dL | 0.6 (5.8) | 0.6 (8.6)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in HDL at Week 4; Test type: Superiority or Other; p = 0.739, ANCOVA — No adjustment for p-value for secondary analyses; difference in LS Means = -0.30, 95% CI [-2.07 to 1.47]

17. Secondary Outcome: Change in Total Cholesterol (TC) From Baseline to Week 4.
Description: Mean change at observation minus baseline.
Time Frame: Week 4, baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mg/dL | 0.5 (23.5) | -55.9 (26.8)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in TC at Week 4; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -57.9, 95% CI [-64.02 to 51.81]

18. Secondary Outcome: Change From Baseline in Triglycerides (TG) to Week 4.
Description: Mean change at observation minus baseline
Time Frame: Week 4, baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mg/dL | 2.4 (73.2) | -45.7 (62.8)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in TG at Week 4; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -47.27, 95% CI [-63.37 to -31.16]

19. Secondary Outcome: Change From Baseline in LDL at Week 6.
Description: Mean change at observation minus baseline.
Time Frame: Week 6, baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mg/dL | 0.3 (24.8) | -49.2 (24.0)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in LDL at Week 6; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -51.21, 95% CI [-56.88 to -45.55]

20. Secondary Outcome: Change From Baseline in HDL at Week 6.
Description: Mean change at observation minus baseline.
Time Frame: Week 6, baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mg/dL | 1.2 (8.2) | 0.4 (8.2)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in HDL at Week 6; Test type: Superiority or Other; p = 0.329, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -1.02, 95% CI [-3.07 to 1.03]

21. Secondary Outcome: Change From Baseline in Total Cholesterol (TC) to Week 6.
Description: Mean change at observation minus baseline.
Time Frame: Week 6, baseline
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mg/dL | 3.7 (23.8) | -56.8 (28.4)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline in TC at Week 6; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -62.07, 95% CI [-68.49 to -55.65]

22. Secondary Outcome: Change From Baseline in Triglycerides (TG) at Week 6.
Description: Mean change at observation minus mean baseline.
Time Frame: Week 6 , baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
mg/dL | 11.6 (115.3) | -42.6 (67.3)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change in TG from baseline in at Week 6; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -53.95, 95% CI [-77.61 to -30.29]

23. Secondary Outcome: Change From Baseline to Week 4 in Framingham Predicted Absolute 10-year Risk.
Description: Framingham prediction of absolute 10-year risk of CHD outcomes (MI or CHD death) are calculations based on total point score (range less than negative 3 [best] to greater than or equal to 14 [worst] for men; less than or equal to negative 2 [best] and greater than or equal to 17 [worst] for women) of subject age, sex, current blood pressure treatment status, current smoking status, total cholesterol, high-density lipoprotein cholesterol and systolic blood pressure calculated at Week 4. Mean at observation minus mean at baseline.
Time Frame: Week 4, baseline
Population: as for outcome 3
Measure: Least Squares Mean (Standard Deviation); unit: score on scale
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
score on scale | -0.3 (2.5) | -2.8 (3.3)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in mean change from baseline to Week 4 in Framingham predicted absolute 10-year risk; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -2.4, 95% CI [-3.1 to -1.7]

24. Primary Outcome: Change From Baseline to Week 6 in Framingham Predicted Absolute 10-year Risk
Description: Framingham prediction of absolute 10-year risk of Coronary Heart Disease (CHD) outcomes (myocardial infarction [MI] or CHD death) are calculations based on total point score (range less than negative 3 [best] to greater than or equal to 14 [worst] for men; less than or equal to negative 2 [best] and greater than or equal to 17 [worst] for women) of subject age, sex, current blood pressure treatment status, current smoking status, total cholesterol, high-density lipoprotein cholesterol, and systolic blood pressure calculated at Week 6. Mean at observation minus mean at baseline.
Time Frame: Week 6, baseline
Population: The full analysis set of all randomized subjects who took at least one dose of study drug and had any post-baseline efficacy assessment
Measure: Least Squares Mean (Standard Deviation); unit: score on scale
Arm/Group | Norvasc + TLC | Caduet + TLC
Number analyzed (Participants) | 115 | 118
score on scale | -0.1 (2.9) | -2.9 (3.0)
Statistical Analysis 1: Comparison: Norvasc + TLC vs Caduet + TLC; Null hypothesis: There is no difference between the two treatment management strategies in the mean change from baseline to Week 6 in Framingham predicted absolute 10-year risk; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustment for p-value for secondary analyses; Difference in LS Means = -2.8, 95% CI [-3.5 to -2.1]

ADVERSE EVENTS:
Arm/Group | Norvasc + TLC | Caduet + TLC
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/122
Other Adverse Events (participants affected / at risk) | 16/122 | 7/122
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Norvasc + TLC (N=122) | Caduet + TLC (N=122)
Oedema peripheral (General disorders) | 8 | 3
Urinary tract infection (Infections and infestations) | 3 | 1
Hypertension (Vascular disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.